CLINICAL TRIAL: NCT04186793
Title: Comparison of Dietary Sugar Reduction Methods
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: Center for Cystic Fibrosis and Airways Disease Research (Unknown)
Responsible Party: Principal Investigator, Miriam Vos, Professor, Emory University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB00115167
Record Dates: First submitted 2019-12-03; First posted 2019-12-05 (Actual); Last update posted 2022-03-25 (Actual); Status verified 2022-03

CONDITIONS: Nonalcoholic Fatty Liver Disease
Keywords: Pediatrics; Obesity; Liver Disease
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Obesity; Liver Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Guided Grocery Shopping (Experimental): Participants in this study arm will receive a guided grocery shopping intervention for four weeks.
  Interventions: Behavioral: Guided Grocery Shopping (GGS)
- Diet Provision Group (Experimental): Participants in this study arm will be provided with a diet low in free sugars. This intervention replaces the habitual diet with a low "free sugars" diet (goal of <3% of total calories).
  Interventions: Other: Diet Provision Group

INTERVENTIONS:
Behavioral: Guided Grocery Shopping (GGS) — The GGS group will be scheduled for 4 weekly sessions to co-shop with the study Registered Dietitian (RD) or clinical research coordinator (CRC). The primary shopper for the household will be required to attend all 4 sessions. The study participant will be required to attend at least 1 session and other family/household members will be encouraged to attend. The weekly sessions will take place at the family's primary grocery store. During each session, the RD will facilitate selection of low free sugar foods and guide the primary shopper on menu planning for a low free sugar diet. In the 4th session, the primary shopper will be asked to shop independently while being observed by the RD/CRC. Prior to checking out, the RD/CRC will approve and/or correct their shopping choices.
  During the follow-up period, all participants will receive diet counseling/support calls from the dietitian and/or research team at Months 2, 4, and 6, following intervention completion.
  Arms: Guided Grocery Shopping
Other: Diet Provision Group — This intervention will be applied to each family and will target foods and beverages that contain free sugars added to food by consumer, cook, or manufacturer, but preserve the family's other food group choices. During the 4 week long intervention, families will be able to choose meals from a list of foods similar to their usual diet. Groceries for each week will be delivered to the family. Each child will be provided with a lunch bag and instructed to bring lunch to school to maintain the study diet.
  Families will have the opportunity to choose from a list of pre-prepared evening meals that are similar to what they consumed before study initiation but without free sugars. The families will be instructed to not eat any food outside of the assigned diet.
  During the follow-up period, all participants will receive diet counseling/support calls from the dietitian and/or research team at Months 2, 4, and 6, following intervention completion.
  Arms: Diet Provision Group

SUMMARY:
This is a two arm, randomized, 4 week study comparing 2 methods of dietary sugar reduction at Emory University and Children's Healthcare of Atlanta. Participants will be non-diabetic children with NAFLD. Two groups of 6 participants will be followed for 4 weeks during the randomized controlled trial followed by a 20 week follow-up extension. One group will receive a guided grocery shopping (GGS) intervention for 4 weeks while the other group will be provided with a low free sugars (<3% total daily) diet.

The goal of this study is to determine if guided grocery shopping (GGS) over 4 weeks is equivalent to complete family diet provision in reducing free sugar intake to <3% of total energy (TE) and if GGS will sustain the dietary change over 6 months.

DETAILED DESCRIPTION:
Nonalcoholic fatty liver disease (NAFLD) is a condition in which abnormal amounts of fat deposit in the liver. This ectopic deposition of triglycerides is metabolically harmful to the liver and is strongly associated with dysregulation of lipid metabolism and insulin resistance. NAFLD is increasing in prevalence in children and now is estimated to affect ~30% of obese children in the U.S. and 6-15% of children across the world. The severity of the disease ranges widely, from mild with increased fat (steatosis) alone to more severe phenotypes of steatosis, inflammation and hepatocyte ballooning (called steatohepatitis) to cirrhosis. While the natural course of pediatric NAFLD is not fully understood, in adults, progression to cirrhosis occurs in about 10%. Diabetes is strongly associated with NAFLD and in children the incidence of prediabetes and diabetes in children with NAFLD is 3 to 5% per year, markedly increases from population estimates of 3.5/cases per 100,000.

Because of the high prevalence of NAFLD, especially among children with obesity, and the increased mortality and morbidity associated with NAFLD, it has become a focus for therapeutic development. In children, there have been several phase 2 clinical trials, but to date there no approved medications for NAFLD. The current standard of care for pediatric NAFLD treatment is healthy diet and exercise. Which "healthy diet" to apply is unknown. Short term evidence in adults supports a variety of approaches including Mediterranean diet, low-fat diet, and low-carbohydrate diet.

For children, there has been a focus on diet quality rather than weight loss. In totality, research demonstrates that consumption of free sugars leads to increased triglycerides, decreased high density lipoprotein cholesterol (HDLc) and increased very low density lipoprotein (VLDL) size, as well as endotoxemia, while reduction of free sugars improves hepatic fat and inflammation.

Complete diet provision is established as an effective research tool to test a diet modification. However, this approach becomes impractical, unsustainable, and expensive when applied across a large multicenter trial. Consequently, less intensive methods would be highly beneficial, if they are equally effective in modifying the diet. Thus, this randomized equivalence pilot study has been designed to test if facilitated grocery shopping will be equivalent to complete diet provision in reducing free sugar consumption to ≤ 3% in children with NAFLD.

This is a 4-week randomized, controlled, outpatient feeding study at Emory University and Children's Healthcare of Atlanta. Participants will be non-diabetic children with NAFLD. Two groups of 6 participants will be followed for 24 weeks. This will include 4 weeks during which the randomized controlled trial will be conducted, followed by a 20 week follow-up. One group will receive the guided grocery shopping (GGS) intervention for 4 weeks while the other group will be provided with a low free sugars (goal of <3% total daily calories) version of their family's habitual diets. Both groups will receive diet/nutrition counseling and support once per week during the intervention period.

ELIGIBILITY:
Inclusion Criteria:

* Clinical history consistent with NAFLD
* Written informed consent from parent or legal guardian
* Written or verbal informed assent from the child
* Currently regularly consumes sugary beverages ( ≥ 2 eight ounce sugar drinks or juice per week)

Exclusion Criteria:

* Participants with a history of health issues that make it unsafe for them to participate in the opinion of the investigators
* History of significant depression
* Diabetes
* Evidence of other chronic liver disease
* Children who are currently enrolled in a clinical trial or who received an investigational study drug or dietary intervention within the past 60 days
* Participants who are not able or willing to comply with the diet protocol or have any other condition that would impede compliance or hinder completion of the study, in the opinion of the investigator
* Families with > 6 individuals

Ages: 8 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 8 (Actual)
Dates: Start 2020-02-06 (Actual); Primary Completion 2021-12-15 (Actual); Study Completion 2021-12-15 (Actual)

PRIMARY OUTCOMES:
Change in Percent of Calories from Free Sugars | Baseline, Week 4, Week 24
  The percent of calories from free sugars in the GGS group will be compared to the diet provision group. Participants will complete a dietary recall covering three 24-hour periods.

SECONDARY OUTCOMES:
Diet compliance | Week 4, Week 24
  Perception of diet compliance difficulty will be assessed qualitatively. Semi-structured interviews will be performed with the participant and their parent/guardian at the end of the study to ascertain their experience during the intervention
Ability to Sustain Diet | Week 4, Week 24
  Perception of the ability to sustain the diet will be assessed qualitatively. Semi-structured interviews will be performed with the participant and their parent/guardian at the end of the study to assess their ability to achieve and maintain a low sugar diet.

CONTACTS AND LOCATIONS:
Overall Officials: Miriam Vos, MD, MSPH, Principal Investigator — Emory University
Locations (2):
- United States (2):
  - Children's Healthcare of Altanta, Atlanta, Georgia
  - Emory University, Atlanta, Georgia

IPD SHARING:
Plan to Share IPD: No